CLINICAL TRIAL: NCT03682133
Title: Practice Variation in Colon Cancer Surgery Care in Older Patients
Brief Title: PreColo Practice Variation
Status: Terminated | Type: Observational
Why Stopped: Retrospective part completed, prospective part response too low
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leading the Change; Zorgverzekaars Nederland (Unknown)
Responsible Party: Sponsor
Other Study IDs: PreColo PV
Record Dates: First submitted 2018-07-24; First posted 2018-09-24 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-05

CONDITIONS: Colon Cancer; Aging; Postoperative Complications
Keywords: Prehabilitation; Preoperative care
MeSH Terms: conditions — Colonic Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehabilitation: The care as given in a participating hospital is according to the local guideline and will not be changed for this study. Whether prehabilitation is applied in a participating hospital is based on a predefined definition of oncological surgical prehabilitation.
- Usual care: Guideline based colon cancer surgery, without prehabilitation.

SUMMARY:
This study will answer the question what the practice variation is (in terms of efficiency) in primary colon surgery on patients of 75 years and above related to the application of different modalities of prehabilitation across the Netherlands.

DETAILED DESCRIPTION:
Rationale: Prehabilitation has shown promising results in orthopedic, cardiothoracic and abdominal surgery. However, there is still a lack of data supporting cost-effectiveness of prehabilitation in colon cancer surgery in older patients. Therefore the Dutch guidelines still restrict prehabilitation for research settings.

Objective: This study will answer the question what the practice variation is (in terms of efficiency) in primary colon surgery on patients of 75 years and above related to the application of different modalities of prehabilitation across the Netherlands. Besides, it will show what service factors (including prehabilitation) determine the technical efficiency of primary colon surgery for these patients of 75 years and above.

Study design: This study is a multicenter observational study based on questionnaires and existing data sources, aimed at including 24 different hospitals, of which structural, process and outcome data related to prehabilitation and colon cancer surgery will be registered.

Study population: Patients aged 75 years and above, 10 per participating hospital, who underwent colon cancer surgery in one of the participating hospitals, where prehabilitation is or is not applied. All patients will be followed with questionnaires focusing on process and outcome measures for the hospital period and three months after discharge.

Intervention: Whether or not the intervention (prehabilitation) is judged as part of daily practice in a participating hospital is based on a predefined definition of oncological surgical prehabilitation. The care as given in a participating hospital is according to the local guideline and will not be changed for this study. According to our definition prehabilitation consists at least of a minimum of 2 weeks exercise therapy and a review of the patients nutritional status at least 2 weeks before surgery.

Usual care: Guideline based colon cancer surgery, without prehabilitation. Main study endpoints: Technical efficiency and service factors that determine this technical efficiency of primary colon cancer surgery. The results will be presented anonymously both for patients and hospitals (so there will not be carried out benchmark analyses per center).

Statistical analysis: Data Envelopment Analysis will be carried out. Factors that might explain variability in technical efficiency will be regressed on bias corrected DEA scores (via truncated regression). Ethical considerations: There will be no change in standard procedures in everyday care. The burden for participants is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and above
* Scheduled for colon cancer surgery

Exclusion Criteria:

* Not receiving surgery
* Hematogenous metastasis
* Pretreatment; chemotherapy or radiotherapy
* Rectal cancer

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Outpatients from the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Technical efficiency measured using Data Envelopment Analysis (DEA) | up to 4 months
  Multiple measurements will be aggregated to arrive at one reported value; technical efficiency. Measurements will be invested care, length of stay, mortality, complication rate and PROMs.
Truncated logistic regression analysis | up to 4 months
  Truncated regression analysis will be performed to identify which explanatory variable(s) predict technical efficiency. Possible explanatory variables will be casemix, yes/ no availability of shared care with geriatrics, yes/no availability of prehabilitation in unimodal or multimodal version, mean volume of older colon cancer patients per practice, propensity score for the frailty of the case mix based on age/sex/disabilities, yes/no availability of laparoscopic colon cancer surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel GM Olde Rikkert, Prof. dr., Principal Investigator — Radboud University Medical Center; Hans HW de Wilt, Prof. dr., Study Chair — Radboud University Medical Center; Thea C Heil, Msc., Principal Investigator — Radboud University Medical Center; Barbara C. van Munster, Dr., Study Chair — Gelre Hospitals; René JF Melis, Dr., Study Chair — Radboud University Medical Center; Huub AA Maas, Dr., Study Chair — ETZ; Peter van Duijvendijk, Dr., Study Chair — Gelre Hospitals
Locations (2):
- Netherlands (2):
  - Gelre ziekenhuizen, Apeldoorn, Gelderland
  - Radboudumc, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: No